CLINICAL TRIAL: NCT04674358
Title: The TRANQUILITY Trial: Multi-Center Randomized, Double-Masked, Parallel Design, Vehicle-Controlled Phase 2/3 Clinical Trial to Assess the Efficacy and Safety of 0.25% Reproxalap Ophthalmic Solution Compared to Vehicle in Subjects With Dry Eye Disease
Brief Title: The TRANQUILITY Trial: Clinical Trial to Assess the Efficacy and Safety in Subjects With Dry Eye Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Aldeyra Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADX-102-DED-019
Record Dates: First submitted 2020-12-14; First posted 2020-12-19 (Actual); Results first posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2023-02

CONDITIONS: Dry Eye; Dry Eye Syndromes
Keywords: reproxalap; ADX-102; Tranquility
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Reproxalap Ophthalmic Solution (0.25%) administered QID over two consecutive days. (Experimental)
  Interventions: Drug: Reproxalap Ophthalmic Solution (0.25%)
- Vehicle Ophthalmic Solution administered over two consecutive days. (Placebo Comparator)
  Interventions: Drug: Vehicle Opthalmic Solution

INTERVENTIONS:
Drug: Reproxalap Ophthalmic Solution (0.25%) — Reproxalap Ophthalmic Solution (0.25%) administered over two consecutive days (Day one pre-dry eye chamber and Day two dry eye chamber assessment).
  Arms: Reproxalap Ophthalmic Solution (0.25%) administered QID over two consecutive days.
Drug: Vehicle Opthalmic Solution — Vehicle Ophthalmic Solution administered over two consecutive days (Day one pre-dry eye chamber and Day two dry eye chamber assessment).
  Arms: Vehicle Ophthalmic Solution administered over two consecutive days.

SUMMARY:
The TRANQUILITY Trial: Multi-Center Randomized, Double-Masked, Parallel Design, Vehicle-Controlled Phase 2/3 Clinical Trial to Assess the Efficacy and Safety of 0.25% Reproxalap Ophthalmic Solution Compared to Vehicle in Subjects with Dry Eye Disease.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age (either gender and any race);
* Reported history of dry eye for at least 6 months prior to Visit 1;
* Reported history of use or desire to use eye drops for dry eye symptoms within 6 months of Visit 1

Exclusion Criteria:

* Clinically significant slit lamp findings at Visit 1 that may include active blepharitis, meibomian gland dysfunction (MGD), lid margin inflammation, or active ocular allergies that require therapeutic treatment, and/or in the opinion of the investigator may interfere with study parameters;
* Diagnosis of an ongoing ocular infection (bacterial, viral, or fungal), or active ocular inflammation at Visit 1;
* Contact lens use within 7 days of Visit 1 or anticipate using contact lenses during the trial;
* Eye drop use within 2 hours of Visit 1;
* Previous laser-assisted in situ keratomileusis (LASIK) surgery within the last 12 months;
* Cyclosporine 0.05% or 0.09% or lifitegrast 5.0% ophthalmic solution use within 90 days of Visit 1;
* Be receiving systemic corticosteroid therapy (not including inhaled corticosteroids) within 14 days of Visit 1 or anticipate such therapy throughout the study period;
* Planned ocular and/or lid surgeries over the study period or any ocular surgery within 6 months of Visit 1;
* Temporary punctal plugs during the study that have not been stable within 30 days of Visit 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 329 (Actual)
Dates: Start 2020-11-21 (Actual); Primary Completion 2021-09-12 (Actual); Study Completion 2021-09-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinical Health, Memphis, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 331 randomized subjects, of which 329 were unique (23 in the initial exploratory cohort and 306 in the main cohort). Two subjects in the main cohort were randomized twice by accident and two subjects were randomized but not dosed, making the safety population 327 subjects. The Safety population is presented in the Participant Flow, Baseline Characteristics, and Adverse Events. Efficacy analysis was conducted on subjects in the main cohort (306 subjects, intent-to-treat population).
Groups:
- Reproxalap Ophthalmic Solution (0.25%): Subjects randomized to reproxalap ophthalmic solution administered seven times over two consecutive days
- Vehicle: Subjects randomized to vehicle ophthalmic solution administered seven times over two consecutive days
Period: Overall Study
Arm/Group | Reproxalap Ophthalmic Solution (0.25%) | Vehicle
Started | 164 | 163
Completed | 162 | 160
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- Reproxalap Ophthalmic Solution (0.25%): Reproxalap ophthalmic solution administered seven times over two consecutive days
- Vehicle: Vehicle ophthalmic solution administered seven times over two consecutive days
- Total: Total of all reporting groups
Arm/Group | Reproxalap Ophthalmic Solution (0.25%) | Vehicle | Total
Number analyzed (Participants) | 164 | 163 | 327
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 87 | 82 | 169
  >=65 years | 77 | 81 | 158
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 120 | 238
  Male | 46 | 43 | 89
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 12 | 22
  Not Hispanic or Latino | 154 | 151 | 305
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 12 | 12 | 24
  Black or African American | 18 | 22 | 40
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  White | 132 | 127 | 259
  Other | 0 | 0 | 0
  Multiple | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 164 | 163 | 327
Iris Color (Right Eye) [Count of Participants; unit: Participants]
  Black | 1 | 4 | 5
  Blue | 48 | 44 | 92
  Brown | 75 | 73 | 148
  Hazel | 24 | 18 | 42
  Green | 14 | 23 | 37
  Gray | 2 | 1 | 3
  Other | 0 | 0 | 0
Iris Color (Left Eye) [Count of Participants; unit: Participants]
  Black | 1 | 4 | 5
  Blue | 48 | 44 | 92
  Brown | 75 | 73 | 148
  Hazel | 24 | 18 | 42
  Green | 14 | 23 | 37
  Gray | 2 | 1 | 3
  Other | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Conjunctival Redness Assessed Over 90 Minutes in the Dry Eye Chamber
Description: Change from baseline comparison of reproxalap to vehicle for conjunctival redness on a 0 to 4 scale ( 0 = normal, 4 = prominent), where a high score means a worse outcome. The intervention was administered bilaterally. The least squares mean (standard error) was derived from mixed model repeated measures for change from baseline included baseline, site, treatment group, and nominal time point as fixed effects.
Time Frame: The efficacy assessment period was assessed during the 90-minute dry eye chamber at Day 2; baseline was Pre-Dose #1 at Day 1.
Population: Intent-to-treat population with observed data only
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Reproxalap Ophthalmic Solution (0.25%): Reproxalap ophthalmic solution administered six times over two consecutive days
- Vehicle: Vehicle ophthalmic solution administered six times over two consecutive days
Arm/Group | Reproxalap Ophthalmic Solution (0.25%) | Vehicle
Number analyzed (Participants) | 153 | 153
units on a scale | 0.185 (0.0233) | 0.156 (0.0229)

2. Secondary Outcome: Schirmer Test Change From Baseline After the First Dose on Day 1
Description: Change from baseline comparison of reproxalap to vehicle for Schirmer test on a millimeter line (0 = none, 35 = maximum), where a shorter length indicates a worse outcome. The least squares mean (standard error) was derived from mixed model repeated measures for change from baseline included baseline and treatment group as fixed effects.
Time Frame: The efficacy assessment period was before and after the final dose on Day 1; baseline was Pre-Dose #1 at Day 1.
Population: Intent-to-treat population with observed data only
Measure: Least Squares Mean (Standard Error); unit: millimeters
Groups:
- Reproxalap Ophthalmic Solution (0.25%): Reproxalap ophthalmic solution administered four times over one day
- Vehicle: Vehicle ophthalmic solution administered four times over one day
Arm/Group | Reproxalap Ophthalmic Solution (0.25%) | Vehicle
Number analyzed (Participants) | 153 | 153
millimeters | 5.9 (0.53) | 3.5 (0.53)

3. Post Hoc Outcome: Conjunctival Redness Assessed Over 90 Minutes in the Dry Eye Chamber Using Computer Automated Grading
Description: Change from baseline comparison of reproxalap to vehicle for conjunctival redness on a 0 to 255 scale ( 0 = none, 255 = maximum), where a high score means a worse outcome. The intervention was administered bilaterally. The least squares mean (standard error) was derived from mixed model repeated measures for change from baseline included baseline, site, treatment group, and nominal time point as fixed effects.
Time Frame: as for outcome 1
Population: Intent-to-treat population with observed data only
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Reproxalap Ophthalmic Solution (0.25%) | Vehicle
Number analyzed (Participants) | 153 | 153
units on a scale | 0.309 (0.2160) | 0.962 (0.2121)

4. Post Hoc Outcome: Number of Subject Eyes That Are Schirmer Test Responders (Eyes 10 Millimeters or More Increase From Baseline)
Description: The number of subject eyes that are schirmer test responders (eyes with 10 millimeters or more increase from baseline) using a millimeter line (0 = none, 35 = maximum), where a shorter length indicates a worse outcome.
Time Frame: Efficacy was assessed after a single dose on Day 1; baseline was assessed approximately two weeks before dosing.
Population: Intent-to-treat population with observed data only
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Reproxalap Ophthalmic Solution (0.25%) | Vehicle
Number analyzed (Participants) | 153 | 153
Number analyzed (eyes) | 306 | 306
eyes | 125 | 64
Statistical Analysis 1: Comparison: Reproxalap Ophthalmic Solution (0.25%); Test type: Superiority; Odds Ratio (OR) = 2.63, 95% CI 2-sided [1.67 to 4.14]

ADVERSE EVENTS:
Time Frame: The period of time over which adverse events were collected for each subject in the clinical trial was approximately one week.
Arm/Group | Reproxalap Ophthalmic Solution (0.25%) | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/164 | 0/163
Serious Adverse Events (participants affected / at risk) | 0/164 | 0/163
Other Adverse Events (participants affected / at risk) | 118/164 | 2/163
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Reproxalap Ophthalmic Solution (0.25%) (N=164) | Vehicle (N=163)
General disorders and administration site conditions (General disorders) | 118 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-11-05): https://cdn.clinicaltrials.gov/large-docs/58/NCT04674358/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-17): https://cdn.clinicaltrials.gov/large-docs/58/NCT04674358/SAP_001.pdf